CLINICAL TRIAL: NCT05640206
Title: Effect of Intra-articular Injection of Injectable Platelet-rich Fibrin on Disc Displacement Without Reduction
Brief Title: Effect of Injectable Platelet-rich Fibrin on Disc Displacement Without Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Assistan Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22038
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Disc Disorder
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): intra-articular i-PRF injection after arthrocentesis
  Interventions: Procedure: i-PRF
- Control group (Experimental): only arthrocentesis
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: i-PRF — Arthrocentesis performed with two-needle technique, and then injection of i-PRF intra-articularly
  Arms: Test group
Procedure: Arthrocentesis — Arthrocentesis performed with two-needle technique
  Arms: Control group

SUMMARY:
This randomized clinical study was conducted on patients with disc displacement without reduction. Patient was selected one of the two study groups: control group received only arthrocentesis or test group received arthrocentesis + injectable platelet-rich fibrin (i-PRF). As primary outcome variable, pain was recorded at preoperatively and at postoperatively 1, 2, 3, 6 and 12 months. Maximum mouth opening, lateral and protrusive movements were formed as secondary outcome variables.

DETAILED DESCRIPTION:
This randomized clinical study was conducted on patients with disc displacement without reduction. Patient was selected one of the two study groups: control group received only arthrocentesis or test group received arthrocentesis + i-PRF. Arthrocentesis procedure was performed for all groups with two needle technique. For test group, intra-articular i-PRF was made. As a primary outcome variable, pain was recorded at preoperatively and at postoperatively 1, 2, 3, 6 and 12 months. Maximum mouth opening, lateral and protrusive movements were formed as secondary outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral disc displacement without reduction
* localized pain on temporomandibular joint
* decreased mouth opening, lateral and protrusive movements

Exclusion Criteria:

* Malignant or inflammatory disorders
* prior surgical history of temporomandibular joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change of pain | at preoperatively, and at 1, 2, 3, 6 and 12 months postoperatively
  Pain was measured with a 10-point visual analogue scale which range from 0 meaning no pain to 10 meaning worst pain at preoperatively and at 1, 2, 3, 6 and 12 months postoperatively

SECONDARY OUTCOMES:
Change of maximum mouth opening | at preoperatively, and at 1, 2, 3, 6 and 12 months postoperatively
  Maximum mouth opening was measured with a millimeter ruler at preoperatively and at 1, 2, 3, 6 and 12 months postoperatively
Change of lateral movements | at preoperatively, and at 1, 2, 3, 6 and 12 months postoperatively
  Lateral movements were measured with a millimeter ruler at preoperatively and at 1, 2, 3, 6 and 12 months postoperatively
Change of protrusive movements | at preoperatively, and at 1, 2, 3, 6 and 12 months postoperatively
  Protrusive movements were measured with a millimeter ruler at preoperatively and at 1, 2, 3, 6 and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Işık, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No